CLINICAL TRIAL: NCT00299221
Title: Tacrolimus In Combination, Tacrolimus Alone Compared (TICTAC Trial): A Prospective Randomized Trial Of Minimized Immunosuppression In Adult Heart Transplant Recipients
Brief Title: Safety Outcomes of Lower Immunosuppression Versus Traditional Immunosuppression in Heart Transplant Recipients
Acronym: TICTAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newark Beth Israel Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, David A. Baran, MD, Director, Heart Failure and Transplant Research, Newark Beth Israel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TICTAC
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Immunosuppression
Keywords: immunosuppression; steroid withdrawal; rejection; coronary disease; cytomegalovirus infection
MeSH Terms: conditions — Rejection, Psychology; Coronary Disease; Cytomegalovirus Infections | interventions — Tacrolimus; Combined Modality Therapy; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy (Active Comparator): Tacrolimus alone
  Interventions: Drug: Tacrolimus
- Combination therapy (Active Comparator): tacrolimus with mycophenolate mofetil
  Interventions: Drug: Tacrolimus; Drug: combination therapy

INTERVENTIONS:
Drug: Tacrolimus — tacrolimus
  Other Names: Prograf
Drug: combination therapy — MMF
  Other Names: mycophenolate mofetil / CellCept
  Arms: Combination therapy

SUMMARY:
This was a study to compare less intense immunosuppression with a more traditional approach. The hypothesis was that less immunosuppression will provide similar protection against rejection than typical 2-3 drug therapy.

DETAILED DESCRIPTION:
This was a prospective, randomized, controlled (open-label) trial of 2 different strategies of immunosuppression in de novo post-heart transplant patients. The hypothesis was that immunosuppression with tacrolimus and mycophenolate mofetil, coupled with rapid steroid weaning would provide similar anti-rejection efficacy as tacrolimus with only a 2 week course of mycophenolate mofetil but including the same rapid steroid wean.

The primary endpoint was the mean International Society for Heart and Lung Transplantation (ISHLT) biopsy score over the first 6 months post-transplant. Secondary endpoints included the incidence of adverse events over the first year post-transplant, as well as all-cause mortality, 12 month ISHLT biopsy score (mean), along with the incidence of proven cytomegalovirus disease. In addition, the incidence of allograft vasculopathy as assessed by angiography or intravascular ultrasound was compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years old)
* Undergoing a first heart transplant (no heart/kidney transplants), who receive their transplant at one of the study sites
* Specifically INCLUDED are patients on ventricular assist devices, and allosensitized recipients

Exclusion Criteria:

* Age less than 18
* Inability to provide proper informed consent
* Combined organ transplantation
* Re-Transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Baran, MD, Principal Investigator — Newark Beth Israel Medical Center
Locations (2):
- United States (2):
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mt. Sinai Cardiovascular Institute, New York, New York

REFERENCES:
- [Result] Baran DA, Zucker MJ, Arroyo LH, Alwarshetty MM, Ramirez MR, Prendergast TW, Goldstein DJ, Camacho M, Gass AL, Carr C, Cohen M. Randomized trial of tacrolimus monotherapy: tacrolimus in combination, tacrolimus alone compared (the TICTAC trial). J Heart Lung Transplant. 2007 Oct;26(10):992-7. doi: 10.1016/j.healun.2007.07.022. PMID 17919618
- [Result] Baran DA, Zucker MJ, Arroyo LH, Camacho M, Goldschmidt ME, Nicholls SJ, Prevost-Fernandez J, Carr C, Adams L, Pardi S, Hou V, Binetti M, McCahill J, Chichetti J, Viloria V, Sanagustin MG, Ebuenga-Smith J, Mele L, Martin A, Blicharz D, Wolski K, Olesnicky L, Qian F, Gass AL, Cohen M. A prospective, randomized trial of single-drug versus dual-drug immunosuppression in heart transplantation: the tacrolimus in combination, tacrolimus alone compared (TICTAC) trial. Circ Heart Fail. 2011 Mar;4(2):129-37. doi: 10.1161/CIRCHEARTFAILURE.110.958520. Epub 2011 Jan 7. PMID 21216835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pts recruited from April 2004-Aug 2008
Pre-assignment Details: Consent often obtained after transplant
Groups:
- Monotherapy: These patients will receive tacrolimus, mycophenolate mofetil (MMF) and corticosteroids, followed by a rapid 8 week wean of steroids to discontinuation. MMF will be discontinued in this group at 14 days post-transplant
- Combination Therapy: These patients will receive tacrolimus, mycophenolate mofetil (MMF) and corticosteroids, followed by a rapid 8 week wean of steroids to discontinuation. MMF will be maintained in this group, unless intolerance develops.
Period: Overall Study
Arm/Group | Monotherapy | Combination Therapy
Started | 79 | 71
Completed | 79 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 79 | 71 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 57 | 121
  >=65 years | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.7) | 54.6 (11.6) | 54.65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 62 | 60 | 122
Region of Enrollment [Number; unit: participants]
  United States | 79 | 71 | 150

OUTCOME MEASURES:

1. Primary Outcome: Mean International Society for Heart and Lung Transplantation Biopsy Score Over the First 6 Months Post-transplantation
Description: Mean ISHLT biopsy score Biopsies of the heart may be various grades and each is assigned a numerical score. Grade 0 is 0 points, 1A = 1, 1B = 2, grade 2 = 3, grade 3A = 4, Grade 3B = 5, and grade 4 = 6 units. The mean biopsy score is the numeric average of the biopsy scores for the first 6 post-transplant months. Best value is 0, worst score is 6.
Time Frame: 6 months
Population: all pts, intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 79 | 71
units on a scale | 0.7 (0.44) | 0.65 (0.4)

2. Secondary Outcome: Percent of Patients Alive at One Year Post-transplant
Description: Percent of patients alive at one year post-transplant. In other words, all cause mortality over time
Time Frame: 1 year
Population: all pts, intention to treat
Measure: Number; unit: percent of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 79 | 71
percent of participants | 98 | 98

3. Secondary Outcome: Number of Patients With Cytomegalovirus (CMV) at One Year Post-transplant
Description: Number of patients developing cytomegalovirus disease by 1 year post-transplant
Time Frame: 1 year
Population: all patients
Measure: Number; unit: participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 79 | 71
participants | 2 | 2

4. Secondary Outcome: Number of Patients With Allograft Vasculopathy (CAD) at One Year Post Transplant
Description: Number of patients diagnosed with allograft vasculopathy / coronary artery disease (CAD) at one year post transplant
Time Frame: 1 year
Population: Percent of patients with allograft CAD at one year post-transplant
Measure: Number; unit: patients
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 79 | 71
patients | 0 | 0

5. Secondary Outcome: Mean ISHLT Biopsy Score Over First Year Post-transplant
Description: as for outcome 1
Time Frame: 1 year
Population: all pts, Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 79 | 71
units on a scale | 0.67 (0.39) | 0.62 (0.39)
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; comparing ISHLT biopsy score between groups at 1 year; Test type: Superiority or Other; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = .2, Standard Deviation .4

ADVERSE EVENTS:
Time Frame: 1 year
Description: Cytomegalovirus (CMV) disease
Arm/Group | Monotherapy | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 2/79 | 1/71
Other Adverse Events (participants affected / at risk) | 0/79 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy (N=79) | Combination Therapy (N=71)
death (General disorders) | 2 (2) | 1 (1) — mortality, tabulated as secondary outcome measure

LIMITATIONS AND CAVEATS:
This trial enrolled 150 patients, but cannot be used to generalize care to other patients without careful consideration of risks and benefits. All patients had corticosteorids weaned so this trial doesn't assess the risk of steroid weaning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No